CLINICAL TRIAL: NCT04783961
Title: Cold Snare Endoscopic Resection for Duodenal Adenomas
Acronym: COLD SNARE
Status: Completed | Type: Observational
Sponsor: Istituto Clinico Humanitas (Other)
Responsible Party: Sponsor
Other Study IDs: 2248
Record Dates: First submitted 2021-03-02; First posted 2021-03-05 (Actual); Last update posted 2022-09-15 (Actual); Status verified 2022-09

CONDITIONS: Duodenal Adenomas

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Cold snare endoscopic resection — Cold snare endoscopic resection

SUMMARY:
Non-ampullary sporadic duodenal adenomas (SDA) are rare lesions, incidentally discovered in up to only 5% of patients during routine endoscopy. In any case, these lesions require treatment due to their potential malignant transformation because of the adenoma-carcinoma sequence, occurring in 30-85% of cases. Endoscopic resection (ER) of SDA represents an attractive alternative to surgical resection in appropriately selected patients, with lower morbidity and mortality rates.

However, most endoscopists are not keen to resect larger lesions due to the risk of complications. Indeed, endoscopic resection in the duodenum has unique challenges: thin wall, high vascularity, very limited space and harmful effects of bile and acid both acting on the ER defect.

Cold snare endoscopic resection has been shown to be a viable method for removing colorectal lesions with comparable efficacy outcomes compared to conventional polypectomy/endoscopic mucosal resection (EMR) and a promising safety profile. As a matter of fact, adverse events associated with hot snare resection technique such as delayed bleeding, post-polypectomy syndrome, and perforation are all related to electrocautery-induced injury.

Performing cold snare piece-meal resection and avoiding the need of thermal therapy, may have a major impact in the duodenum where the risk of delayed bleeding and perforation is consistent.

The aim of this pilot study is to prospectively evaluate the feasibility and the efficacy in term of safety and efficacy of cold snare endoscopic resection.

ELIGIBILITY:
Inclusion Criteria:

• Patients able to give informed consent to involvement in trial.

Exclusion Criteria:

* Patient's with known strictures/stenosis
* Pregnancy
* Patients who did not consent to study
* Bleeding diathesis
* Anticoagulants

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with diagnosed large duodenal adenomas (>20 mm)
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Number of patints that will have serious and non-serious adverse events | 3 Months
  * endoscopic appearance
  * scar biopsies
  * perforation risk
Number of residual adenomas | 3 Months
  * endoscopic appearance
  * scar biopsies

SECONDARY OUTCOMES:
Duration of endoscopic procedure | 3 Months
Hospital stay | 3 Months
Hospital readmission | 3 Months

CONTACTS AND LOCATIONS:
Locations (1):
- Endoscopy Unit, Humanitas Research Hospital, Rozzano, Milano, Italy

IPD SHARING:
Plan to Share IPD: No